CLINICAL TRIAL: NCT03637582
Title: Contribution of Urethral Sensory Feedback in Voiding Efficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00071589_1
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-01

CONDITIONS: Urethral Anesthesia
Keywords: voiding efficiency; detrusor underactivity; urodynamics
MeSH Terms: conditions — Urinary Bladder, Underactive | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anesthesia Arm (Active Comparator): Participants randomized to this arm will undergo uroflow studies then be given an hour rest. Five ml of 4% lidocaine gel will be inserted into the urethra during their hour rest. After the incubation period, the subject will receive another five ml of 4% lidocaine gel. The subject will then perform the second uroflow study.
  Complex urodynamics with the use of lidocaine hydrochloride 4% will then be performed. The lidocaine gel will have been placed in and around the urethra. We are using lidocaine gel in an FDA approved manner (for anesthesia).
  Interventions: Drug: lidocaine gel
- Placebo Arm (Placebo Comparator): Participants randomized to this arm will first undergo uroflow studies then be given an hour rest. Five ml of plain aqueous gel will be inserted into the urethra during their hour rest. After the incubation period, the subject will receive another five ml of plain aqueous gel. Urodynamic testing without anesthesia (standard of care) will then be performed.
  Interventions: Other: Plain aqueous gel

INTERVENTIONS:
Drug: lidocaine gel — Lidocaine (4%) gel from Quest Products, Inc.
  Other Names: 4% lidocaine
  Arms: Anesthesia Arm
Other: Plain aqueous gel — KY jelly lubricant from Reckitt Benckiser
  Other Names: KY gel
  Arms: Placebo Arm

SUMMARY:
The purpose of this study is to evaluate how urethral anesthesia impacts voiding efficiency in healthy women. The investigator hypothesizes that anesthetizing the urethral with lidocaine gel will decrease voiding efficiency as measured by standard bladder testing (urodynamic testing).

DETAILED DESCRIPTION:
1. Purpose of the Study

   The purpose of this study is to determine whether urethral sensory feedback has a role in the micturition (bladder emptying) reflex in female controls during routine office Urodynamic Studies (UDS). UDS are current clinical tests of urethral and bladder function and consist of several individual studies including filling cystometry, pressure-flow studies, and urethral pressure profilometry (UPP). Filling cystometry focuses primarily on sensation and activity of the bladder during the filling (or storage) phase of the micturition (voiding) cycle. Pressure-flow studies (which include voiding cystometry) are used to assess the motor activity of the bladder muscle during bladder emptying. UPP assesses urethral sphincter motor function and has traditionally been used to evaluate stress urinary incontinence. Perineal patch electromyography (EMG) is often added to UDS to assess for pelvic floor muscle recruitment during voiding, which may suggest voiding dysfunction.
2. Background & Significance

   The storage and elimination of urine is regulated by neural circuits in the brain and spinal cord to coordinate function between the urinary bladder and the urethra (Fowler, Griffiths et al. 2008). During the micturition (bladder emptying) reflex, the elimination of urine is facilitated by bladder wall contraction and urethral wall and pelvic floor muscle relaxation. Urine that subsequently flows through the urethra also activates sensory nerves to amplify bladder contractions and maintain efficient bladder emptying (Jung, Fraser et al. 1999, Bump 2000). Incomplete voiding and urinary retention occurs when these mechanisms are disrupted or poorly coordinated.

   Incomplete bladder emptying due to detrusor underactivity is an understudied health concern for women in the United States. The overall incidence of detrusor underactivity in women has not yet been reported in the literature. One study by Wu et al. (2005) determined that 7.8% of patients in an outpatient rehabilitation facility had symptoms of incomplete bladder emptying; whereas, 21% of people without symptoms had elevated post void residuals when universally screened. Their population consisted of 350 patients, of which two-thirds were women. Lower urinary tract symptoms, including urinary urgency, frequency and incomplete bladder emptying, have been shown to decrease quality of life, increase healthcare utilization, decrease workplace productivity, and impact intimate relationships (Richter et al. 2007, Coyne et al. 2003).

   The current clinical management options for women with retention are intermittent or indwelling catheterization, urethral dilation, or reconstructive surgery (Mevcha and Drake 2010). These treatments, however, often fail to completely resolve lower urinary tract symptoms and the patients may develop chronic retention complications such as overflow incontinence, hydroureter, hydronephrosis, infection, or renal failure. In order to improve therapeutic outcomes, there is still a need to clarify the specific mechanisms that underlie detrusor underactivity in women. Our proposed studies will be contributing to the growing body of literature implicating urethral sensory feedback as a candidate to recover efficient bladder emptying.
3. Hypothesis and Justification

   Overall Hypothesis: Urethral afferent nerve fiber activation augments bladder contractions for efficient voiding and urethral anesthesia will disrupt sensory feedback and impair bladder emptying.

   Specific Aim 1: To assess voiding efficiency (voided volume/{voided volume + residual volume}) in women controls with and without urethral anesthesia.

   Hypothesis 1a: Voiding efficiency will be lower when the urethra is anesthetized during uroflow studies

   Hypothesis 1b: Detrusor contraction at maximum flow rate (Pdet@Qmax) and duration of detrusor contraction will be reduced when the urethra is anesthetized during micturition pressure-flow studies

   Hypothesis 1c: Voiding while anesthetized will lead to increased valsalva-voiding (increased intra-abdominal pressure, Pabd) and an intermittent urinary stream during micturition pressure-flow studies

   Specific Aim 2: To assess whether urethral anesthesia gel improves discomfort during the UDS

   Hypothesis 2a: Visual Analog Scale (VAS) scores for pain will be lower during the UDS when the urethra has been anesthetized
4. Studies Supporting Specific Aims:

   i. Micturition with Urethral Anesthesia: Distension and fluid flow in the urethra has been previously demonstrated to evoke sensory nerve discharge. Nerve firing originating from the urethra is then able to initiate contractions in the filling bladder and increase the amplitude and duration of ongoing bladder contractions. This pudendal-bladder reflex has been shown to be necessary for efficient bladder emptying because disruption to urethral sensory feedback by transection of the sensory branch of the pudendal nerve or intraurethral anesthesia reduces voiding efficiency in the rat. Urethral anesthesia in humans has also been demonstrated to increase post void residual and alter symptoms experienced during the voiding phase.

   This investigator's approach is novel as this study will characterize voiding in healthy women who will be randomized to placebo versus urethral anesthesia. Investigators will do this by performing UDS, which will include all clinical tests for bladder function, with or without urethral anesthesia (4% lidocaine hydrochloride gel or plain aqueous gel).

   ii. Pain Perception During Catheterization: Urethral catheterization elicits mild to moderate pain in women. The use of lubricant anesthetic on the catheter is one available option to manage tissue trauma and pain perception. Several studies have reported that 4% lidocaine gel reduces procedural pain during female urethral catheterization. Others however, have found that lubricant anesthetic and catheter size, does not effect the perception of pain in urethral catheterization in women. These discrepant reports suggest a consensus has not been reached on the efficacy of lubricant anesthetic and pain perception in women.
5. Subject Recruitment: Subjects will be recruited from Duke Hospital and Duke University Campus via newspaper advertisements and paper fliers.
6. Design and Procedures: To account for screen failures, it is anticipated that a total of 30 female controls will be screened to achieve n=20 for completed UDS. Participants will be randomized to their arm of the study using a random number generator. Study staff and the subjects will be blinded to the treatment regimen; thus, our study design is a randomized double-blind placebo-controlled trial.

Study Visit Questionnaires and Tests: After their phone screen, participants will be scheduled for the study visit. All study procedures will take place at the Duke Urogynecology Office at Patterson Place. Participants will undergo informed consent on arrival to their study visit. They will provide a urine specimen for a point of care urinalysis and pregnancy test. Pre-procedure vital signs, including height and weight will be obtained. They will fill out the following questionnaires: Lower Urinary Tract Symptoms Tool, Sociodemographics and Functional Comorbidity Index and complete a Medication List.

If subjects have a negative urinalysis and pregnancy test they will undergo examination to ensure no evidence of pelvic organ prolapse. A baseline uroflow study will then be performed. The subject will be instructed to void on a commode chair. A post void residual urine measurement will be performed via a bladder scanner. The subject will then complete a baseline VAS. Provided the subject has a normal baseline uroflow and no reported pain on baseline VAS, the subject will be randomized to an arm (lidocaine or aqueous gel first) of the urodynamic study. If either of their point of care tests is positive (per exclusion criteria), they will be excluded from the study and referred to their primary care physician.

Prior to performing UDS, the subject's bladder will be scanned transabdominally with a standard clinic bladder scanner. This will ensure adequate urine is within the bladder prior to beginning. If the subject has > 250mL and < 650mL in their bladder, they will proceed to the UDS procedure room. If the subject has < 250 mL, they will be given a bottle of water and will return to the waiting room for 15-30 minutes. Adequate urine volume will again be confirmed via bladder scanning. Urodynamic testing will then begin.

Order of Studies Performed During Urodynamic Testing: Complex Uroflowmetry, Complex Cystometry, Urethral Pressure Profilometry, Micturition Pressure-flow Study

The Visual Analog Scale (VAS) will be administered to assess discomfort at the following times; after uroflow but before PVR (for baseline and the second study condition uroflow), immediately after the urethral catheter is placed, after 100mL of fluid has been instilled, and at full bladder capacity (MCC).

After the completion of both UDS procedures, participants will be given standard Urogynecology post urodynamics instructions.

ELIGIBILITY:
Inclusion Criteria:

* Females ages 18-60 years
* No health conditions as indicated in exclusion criteria
* Able to provide informed consent and agree to the risks of the study
* Willing to abstain from caffeine and alcohol for 24 hours
* Willing to avoid taking anticholinergic medications (for reasons other than incontinence; e.g., diphenhydramine) for one week prior to the procedure

Exclusion Criteria:

* Pelvic organ prolapse past the hymen
* Multiple sclerosis, myasthenia gravis, Parkinson's Disease, stroke within the past 6 months
* Interstitial cystitis / Bladder Pain Syndrome
* Recurrent (≥ 3/year) urinary tract infections
* Positive pregnancy test at the time of consent
* Positive urine dip (>+1nitrites or >1+LE) and urinary symptoms at the time of consent
* >1+ blood on urinary dip
* Morbid obesity (BMI >40)
* Taking anticholinergic medications for urinary incontinence
* >2 replies of ≥ "sometimes" on the Lower Urinary Tract Symptoms questionnaire at the time of consent
* Alcoholism or failed CAGE questionnaire
* Abnormal baseline uroflow
* Reported pain on baseline VAS (score >10)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Voiding Efficiency | duration of urodynamic study, 2 hours
  voided volume/{voided volume + residual volume} during micturition study during urodynamic studies

SECONDARY OUTCOMES:
Detrusor pressure at maximum flow | duration of urodynamic study, 2 hours
  bladder pressure reading (mmHg) during maximum flow during micturition
Presence or absence of voiding dysfunction | duration of urodynamic study, 2 hours
  presence of interrupted flow during micturition or valsalva voiding as measured by an increases in abdominal pressure (increase in Pabd catheter reading)
Visual analog scale scores | duration of urodynamic study, 2 hours
  The Visual Analog Scale will measure discomfort during urodynamic studies (total range 1-100). The scale goes from no pain (1) to intolerable pain (100) with higher values representing worse pain.

CONTACTS AND LOCATIONS:
Overall Officials: Warren M Grill, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Campus, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen SC, Grill WM, Fan WJ, Kou YR, Lin YS, Lai CH, Peng CW. Bilateral pudendal afferent stimulation improves bladder emptying in rats with urinary retention. BJU Int. 2012 Apr;109(7):1051-8. doi: 10.1111/j.1464-410X.2011.10526.x. Epub 2011 Aug 23. PMID 21883860
- [Background] Peng CW, Chen JJ, Cheng CL, Grill WM. Improved bladder emptying in urinary retention by electrical stimulation of pudendal afferents. J Neural Eng. 2008 Jun;5(2):144-54. doi: 10.1088/1741-2560/5/2/005. Epub 2008 Apr 22. PMID 18430976
- [Background] Shafik A, Shafik AA, El-Sibai O, Ahmed I. Role of positive urethrovesical feedback in vesical evacuation. The concept of a second micturition reflex: the urethrovesical reflex. World J Urol. 2003 Aug;21(3):167-70. doi: 10.1007/s00345-003-0340-5. Epub 2003 Jul 25. PMID 12898170
- [Background] Kisby CK, Gonzalez EJ, Visco AG, Amundsen CL, Grill WM. Randomized Controlled Trial to Assess the Impact of Intraurethral Lidocaine on Urodynamic Voiding Parameters. Female Pelvic Med Reconstr Surg. 2019 Jul/Aug;25(4):265-270. doi: 10.1097/SPV.0000000000000544. PMID 29300256
- [Result] McKee DC, Gonzalez EJ, Amundsen CL, Grill WM. Randomized Controlled Trial to Assess the Impact of High Concentration Intraurethral Lidocaine on Urodynamic Voiding Parameters. Urology. 2019 Nov;133:72-77. doi: 10.1016/j.urology.2019.08.020. Epub 2019 Aug 26. PMID 31465791